CLINICAL TRIAL: NCT03121326
Title: The Study of Sarcopenia and Aging Biomarkers by the Metabolomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Sponsor
Other Study IDs: 201700245B0
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-03

CONDITIONS: Sarcopenia; Aging
Keywords: Sarcopenia; Aging; Biomarkers; Metabolomics
MeSH Terms: conditions — Sarcopenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood and urine sampling — Ten mL blood and 15mL urine are collected.

SUMMARY:
With the rapid growth of the global elderly population, the studies of the biomarkers of the sarcopenia and aging are under investigation in different ways. The investigators use Metabolomics to explore the biomarkers of the sarcopenia and aging of the senior adults.

DETAILED DESCRIPTION:
Metabolomics is the emerging platform technology to address the complexity of a living system. In translational research, metabolomics approaches may enable the detection of multiple disease risk factors and interactions, disease progression, and response of patients to a particular therapy with or without side effects. Metabolomics may provide comprehensive information and improve diagnosis and prognosis which are particularly promising in human complex degenerative diseases. The investigators use Metabolomics to explore the biomarkers of the sarcopenia and aging of the senior adults.

ELIGIBILITY:
Inclusion Criteria:

* residents of the Chang Gung Health and Culture Village
* mostly independent and do not require nursing assistance
* capable of managing their daily living activities
* aged ≧ 60

Exclusion Criteria:

* None.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 650 residents of the Chang Gung Health and Culture Village aged over 60.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
The biomarkers of the sarcopenia and aging in senior adults. | one year
  Metabolomics to explore the biomarkers of the sarcopenia and aging.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ming Lin, M.D., Study Chair — Chang Gung Memorial Hospital; Mei-Ling Cheng, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided